CLINICAL TRIAL: NCT00356642
Title: A Randomised, Single-Blind, Dose-Rising Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Ten Day Repeat Topical Applications of GW842470X Cream on the Skin of Patients With Atopic Dermatitis
Brief Title: Study Of Single And Ten Day Repeat Atopical Applications Of GW842470X Cream On The Skin Of Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: TPD102031
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Dermatitis, Atopic
Keywords: PK; GW842470X; safety; tolerability; PD; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

ARMS (4):
- Single dose 1 cohort (Experimental): Subjects with body surface area (BSA) disease involvement between 10 and 15% will be included. Subjects will receive either 100 milligrams (mg) GW842470X or placebo in a ratio of 2:1.
  Interventions: Drug: GW842470X; Drug: Placebo
- Repeat dose 1 cohort (Experimental): Subjects with BSA disease involvement between 10 and 15% will be included. Subjects will receive either 100-150 mg GW842470X or placebo in a ratio of 3:1
  Interventions: Drug: GW842470X; Drug: Placebo
- Repeat dose 2 cohort (Experimental): Subjects with BSA disease involvement between 30 and 40% will be included. Subjects will receive either 300-400 mg GW842470X or placebo in a ratio of 3:1
  Interventions: Drug: GW842470X; Drug: Placebo
- Repeat dose 3 cohort (Experimental): Subjects with BSA disease involvement >=50% will be included. Subjects will receive either 500-1000 mg GW842470X or placebo in a ratio of 2:1
  Interventions: Drug: GW842470X; Drug: Placebo

INTERVENTIONS:
Drug: GW842470X — GW842470X will be available as a yellow smooth water-in-oil cream.
Drug: Placebo — GW842470X matching placebo will be available as a yellow smooth water-in-oil cream.

SUMMARY:
The purpose of this study of this study is to investigate the safety, tolerability and pharmacokinetics of GW842470X in patients with atopic dermatitis. GW842470X is an inhibitor of phosphodiesterase 4 (PDE4).

ELIGIBILITY:
Inclusion criteria:

* Atopic dermatitis patients (moderate to severe) who are otherwise healthy.
* BMI range 18.5-29.9m2 at least 2 index lesions and BSA involvement >10%.
* 14 day washout of current therapy.

Exclusion criteria:

* Patients who have had systemic treatment for atopic dermatitis or other topical or transdermal treatments (such as nicotine, hormone replacement therapies) within 14 days prior to first application of study medication and/or topical treatment with tar or any treatment with corticosteroids within 14 days prior to first application except 1% hydrocortisone.
* Patients must not present with any systemic disorders or active skin disease other than atopic dermatitis.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-06-10 (Actual); Primary Completion 2005-12-21 (Actual); Study Completion 2005-12-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal physical examination findings | Up to Day 22
Number of subjects with abnormal blood pressure | Up to Day 22
Number of subjects with abnormal heart rate | Up to Day 22
Number of subjects with abnormal 12-lead ECG assessment | Up to Day 22
Number of subjects with abnormal findings on lead II cardiac monitoring | Up to Day 10
Number of subjects with abnormal clinical laboratory tests | Up to Day 22
AUC | Pre-dose, 1, 2, 4, 6, 8, 12 hours on Day 1, pre-dose on Days 3, 5, 7, 9 and pre-dose, 1, 2, 4, 6, 8, 12 , 24, 36 and 48 hours post-dose on Day 10
Cmax | Pre-dose, 1, 2, 4, 6, 8, 12 hours on Day 1, pre-dose on Days 3, 5, 7, 9 and pre-dose, 1, 2, 4, 6, 8, 12 , 24, 36 and 48 hours post-dose on Day 10

SECONDARY OUTCOMES:
Time to max concentration and terminal half-life | Pre-dose, 1, 2, 4, 6, 8, 12 hours on Day 1, pre-dose on Days 3, 5, 7, 9 and pre-dose, 1, 2, 4, 6, 8, 12 , 24, 36 and 48 hours post-dose on Day 10
SCORAD | Up to Day 10
BSA determination | Up to Day 10
clinical photography | Up to Day 10
measurement of barrier function using trans-epidermal water loss (TEWL) | Up to Day 10
skin biopsy (biomarkers CD4+, CD8+, eosinophils, total IgE) | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Ishikawa N, Hattori N, Kohno N, Kobayashi A, Hayamizu T, Johnson M. Airway inflammation in Japanese COPD patients compared with smoking and nonsmoking controls. Int J Chron Obstruct Pulmon Dis. 2015 Jan 23;10:185-92. doi: 10.2147/COPD.S74557. eCollection 2015. PMID 25670894
- See also: Results for study 102031 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/TPD102031?search=study&search_terms=102031#rs